CLINICAL TRIAL: NCT06942845
Title: Exploration of Risk Factors for Postoperative Cerebral Infarction in Lung Cancer Patients: a Retrospective Single-centre Study
Status: Active, not recruiting | Type: Observational
Sponsor: Xinghua Cheng (Other)
Responsible Party: Sponsor-Investigator, Xinghua Cheng, deputy chief physician, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Other Study IDs: postoperative cerebral infarct
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer, Non-Small Cell; Postoperative Cerebral Infarction
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative cerebral infarction
  Interventions: Other: non-intervention
- No postoperative cerebral infarction
  Interventions: Other: non-intervention

INTERVENTIONS:
Other: non-intervention — non-intervention

SUMMARY:
Lung cancer remains the world's leading cancer in terms of morbidity and mortality, with more than 20 million new cases and 9.7 million deaths annually. Despite improvements in surgical techniques and medical care, the number of elderly people undergoing surgery is gradually increasing, so there are an increasing number of complications following lung resection. Postoperative cerebral infarction is a relatively rare but devastating complication that places a heavy burden on patients and families. The incidence of postoperative cerebral infarction in patients after thoracic surgery has been reported to be 0.6-1.1%. There is a risk of postoperative cerebral infarction after lung cancer surgery, and the results of a few studies have shown that postoperative cerebral infarction is related to old age, male, hypertension, hyperlipidemia, and lobectomy factors, but the pathogenesis of the occurrence of cerebral infarction has not been clearly proved for the time being, and so these risk factors cannot be taken as the direct cause of cerebral infarction. Therefore, we need to further explore the factors leading to cerebral infarction after lung cancer surgery. If we can further prove that some of the risk factors are related to the causes of cerebral infarction after lung cancer surgery, we can make corresponding strategies in the perioperative period to improve the safety of surgery and reduce the incidence of cerebral infarction in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

Postoperative cerebral infarction

Exclusion Criteria:

No postoperative infarction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. patients with postoperative cerebral infarction in the hospital during the same period of time as the case group
  2. hospitalised surgical patients in the same period as the control group.
  3. patients who underwent pneumonectomy for lung nodules as the reason for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Analysing independent risk factors for cerebral infarction after pneumonectomy | 5min
  Clinical trial data were entered into Excel for recording information and subsequently converted to SPSS for statistical analysis. Descriptive statistics of the named data were expressed as absolute numbers and percentages according to each patient.
  Clinical characteristics of patients who developed cerebral infarction after surgery were retrospectively compared with those of patients who underwent pneumonectomy without cerebral infarction. Continuous data were expressed as median and interquartile range, and categorical data were expressed as frequencies and percentages. Independent risk factors for developing cerebral infarction after pneumonectomy were analysed using univariate and multivariate logistic regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nishizawa N, Okawara M, Mori M, Fujino Y, Matsuda S, Fushimi K, Tanaka F. Postoperative cerebral infarction risk is related to lobectomy site in lung cancer: a retrospective cohort study of nationwide data in Japan. BMJ Open Respir Res. 2022 Jul;9(1):e001327. doi: 10.1136/bmjresp-2022-001327. PMID 35868837
- [Background] Matsumoto K, Sato S, Okumura M, Niwa H, Hida Y, Kaga K, Date H, Nakajima J, Usuda J, Suzuki M, Souma T, Tsuchida M, Miyata Y, Nagayasu T. Frequency of cerebral infarction after pulmonary resection: a multicenter, retrospective study in Japan. Surg Today. 2018 May;48(5):571-572. doi: 10.1007/s00595-017-1620-9. Epub 2018 Jan 11. No abstract available. PMID 29327086
- [Background] Gao S, Zhou Y, Yang R, Du C, Wu Y. Risk factors for postoperative cerebral infarction in patients after lung resection: a single-center case-control study. J Thorac Dis. 2023 Feb 28;15(2):376-385. doi: 10.21037/jtd-22-1019. Epub 2023 Jan 16. PMID 36910048
- [Background] Hattori A, Takamochi K, Kitamura Y, Matsunaga T, Suzuki K, Oh S, Suzuki K. Risk factor analysis of cerebral infarction and clinicopathological characteristics of left upper pulmonary vein stump thrombus after lobectomy. Gen Thorac Cardiovasc Surg. 2019 Feb;67(2):247-253. doi: 10.1007/s11748-018-1017-8. Epub 2018 Sep 24. PMID 30251002
- [Background] Nojiri T, Inoue M, Takeuchi Y, Maeda H, Shintani Y, Sawabata N, Hamasaki T, Okumura M. Impact of cardiopulmonary complications of lung cancer surgery on long-term outcomes. Surg Today. 2015 Jun;45(6):740-5. doi: 10.1007/s00595-014-1032-z. Epub 2014 Sep 19. PMID 25236860